CLINICAL TRIAL: NCT02462408
Title: A Prospective, Randomized Comparison Between Lateral and Posterior Approach In Ultrasound-Guided Parasagittal In-Plane Infraclavicular Brachial Plexus Block
Brief Title: Conventional Versus Posterior Approach in Ultrasound-Guided Parasagittal In-Plane Infraclavicular Brachial Plexus Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Beh Zhi Yuen, Anaesthetist, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 949.14
Record Dates: First submitted 2015-04-01; First posted 2015-06-04 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Brachial Plexus Block; Infraclavicular; Ultrasound Guided

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Posterior approach (Experimental): The main difference between this block approach and the conventional infraclavicular approach is the site and angle of needle insertion. Otherwise, the end point of local anaesthetic injection remained the same for both approaches.
  Interventions: Procedure: Posterior approach
- Conventional approach (Active Comparator): The main difference between this block approach and the conventional infraclavicular approach is the site and angle of needle insertion. Otherwise, the end point of local anaesthetic injection remained the same for both approaches.
  Interventions: Procedure: Conventional approach

INTERVENTIONS:
Procedure: Posterior approach — The needle insertion point was over the trapezius muscle sufficiently posterior to allow the needle to pass between the clavicle and the scapula in the direction of the axillary artery. The insertion point was strictly aligned with the long axis of the ultrasound beam i.e. in-plane technique.
  Arms: Posterior approach
Procedure: Conventional approach — The needle insertion point would be at the cephalad (lateral) aspect of the ultrasound probe, beneath the clavicle and medial to the coracoid process. The insertion point was strictly aligned with the long axis of the ultrasound beam i.e. in-plane technique.
  Arms: Conventional approach

SUMMARY:
The lateral parasagittal in-plane is the current conventional approach in ultrasound-guided infraclavicular brachial plexus block. However this technique is less popular because brachial plexus at the infraclavicular level runs deeper compared to its course proximally, often give rise to impaired needle visualisation due to its steep angle of needle trajectory to the ultrasound beam. A new posterior parasagittal in-plane approach was introduced to improve needle visibility. This approach proved feasible from our case series hence the investigators would like to compare it with the conventional method in this study

DETAILED DESCRIPTION:
This study compared the conventional lateral and posterior approach parasagittal in-plane ultrasound guided infraclavicular brachial plexus block for upper limb surgery. A cadaveric study was also performed to complement the findings.

After obtaining approval from the Medical Ethics Committee, University Malaya Medical Centre (IRB reference no. 949.14 dated 17 October 2012), 46 patients undergoing upper limb surgery were prospectively recruited and randomized. A cadaveric dissection was also performed.

DESIGN: Prospective randomized study

SETTING: Single centre, University of Malaya Medical Centre, Kuala Lumpur, Malaysia; November 2012 to October 2013

INTERVENTION: Ultrasound guided, lateral or posterior parasagittal in-plane infraclavicular brachial plexus blocks were performed on patients, depending on randomization. All blocks were performed using 21G x 4 inch Stimuplex A (B Braun Medical) without nerve stimulation plus SonoSite M-Turbo with HFL38x/ 13-6 MHz linear transducer probe. A 25-ml local anaesthetic admixture [Lignocaine 2% (100mg) plus Ropivacaine 0.75% (150mg)] were injected to all patients. A total volume of normal saline 0.9% 25ml mixed with methylene blue (0.2ml) was used for cadaveric study.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I - III
* Body Mass Index (BMI) between 20 and 35 kg/m2
* Surgery of the forearm, wrist, or hand

Exclusion Criteria:

* Inability to give consent to the study
* Pre-existing neuropathy
* Infection at the site of puncture, skin ulcer
* Coagulopathy
* Contralateral phrenic nerve paralysis, contralateral recurrent laryngeal nerve paralysis or pneumothorax
* Allergy to amides local anaesthetics

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2012-11; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Success rate (ability to proceed with surgery without the need for intravenous narcotics, general anaesthesia, rescue blocks or local infiltration by the surgeon) | participants will be followed up throughout the operation duration; as stated each operation has variable duration of operation time, average operation time 2 to 4 hours
  Success rate - was equivalent to surgical anesthesia, defined as the ability to proceed with surgery without the need for intravenous narcotics, general anaesthesia, rescue blocks or local infiltration by the surgeon.
  The adequacy of block was determined during assessment of motor and sensory blockade at predetermined intervals, every 5 minutes until 30 minutes; Please refer to the study detailed description.

SECONDARY OUTCOMES:
Performance parameters | participants will be followed up throughout the procedure (performing the blocks), average time for block perfomances 30 minutes
  This is a composite outcome measure. The anaesthesia assistant would record the time required to perform the procedure as follow below description:
  (i)Imaging time (defined as the time interval between contact of the ultrasound probe with the patient and the acquisition of a satisfactory sonoanatomy - a complete round short-axis view of the axillary artery), (ii) Needling time (defined as the time interval between the start of the needle insertion and the end of local anaesthetic injection through the needle), (iii) Performance time (defined as the sum of imaging and needling times). This timing definition had been published in other journals (please refer our references - 3)
Safety aspects and potential complications; we measured by any incidence of paraesthesia, vascular puncture, Horner's syndrome, dyspnoea and symptoms suggestive of LA toxicity | Participants would be followed up throughout procedure (average duration 30 minutes), during operation (average duration 2 to 4 hours) and 1 week after the operation (via phone call)
  This is a composite outcome measure. We measured safety aspects and potential complications by recording any incidence of paraesthesia and vascular puncture during block performances, any Horner's syndrome, dyspnoea and symptoms suggestive of local anaesthetic toxicity were routinely checked after the procedure and during surgery. To further enhance patient's safety, we would still follow up patient by phone call 1 week after the surgery
adequacy of block for tourniquet application | participants would be followed up throughout the operation duration whether they complained of pain at torniquet site during the operation duration; average duration of operation 2 - 4 hours
  The incidence of tourniquet pain; this would describe whether the block technique covers for tourniquet pain

CONTACTS AND LOCATIONS:
Overall Officials: Beh Zhi Yuen, MD, M.Anaes, Principal Investigator — University of Malaya

REFERENCES:
- [Background] Chin KJ, Perlas A, Chan VW, Brull R. Needle visualization in ultrasound-guided regional anesthesia: challenges and solutions. Reg Anesth Pain Med. 2008 Nov-Dec;33(6):532-44. doi: 10.1016/j.rapm.2008.06.002. PMID 19258968
- [Background] Hebbard P, Royse C. Ultrasound guided posterior approach to the infraclavicular brachial plexus. Anaesthesia. 2007 May;62(5):539. doi: 10.1111/j.1365-2044.2007.05066.x. No abstract available. PMID 17448088
- [Background] Tran DQ, Charghi R, Finlayson RJ. The "double bubble" sign for successful infraclavicular brachial plexus blockade. Anesth Analg. 2006 Oct;103(4):1048-9. doi: 10.1213/01.ane.0000239077.49794.a5. No abstract available. PMID 17000840
- [Background] Tran DQ, Bertini P, Zaouter C, Munoz L, Finlayson RJ. A prospective, randomized comparison between single- and double-injection ultrasound-guided infraclavicular brachial plexus block. Reg Anesth Pain Med. 2010 Jan-Feb;35(1):16-21. doi: 10.1097/AAP.0b013e3181c7717c. PMID 20048654